CLINICAL TRIAL: NCT04089527
Title: A Phase 1B Dose Escalation, Multicenter, Open-label Study to Evaluate the Safety, Tolerability, Pharmacokinetic and Pharmacodynamic of CC-95775 in Subjects With Advanced Solid Tumors and Relapsed/Refractory Non-hodgkin's Lymphoma
Brief Title: Study to Evaluate the Safety, Tolerability, Pharmacokinetic and Pharmacodynamic of CC-95775 in Subjects With Advanced Solid Tumors and Relapsed/Refractory Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-95775-ST-001; U1111-1238-6062 (Other: WHO); 2019-001092-36 (EudraCT Number)
Record Dates: First submitted 2019-09-12; First posted 2019-09-13 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: Lymphoma; Non-Hodgkin's Lymphoma; CC-95775; Solid Tumors; Safety; Relapsed/Refractory
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- CC-95775 (Experimental): Escalating dose finding part A of study and extension Part B of the study. In Part A, subjects will be treated with oral capsules of CC-95775 with a schedule of 4d on/ 24d off (Q4W) and a starting dose of 100 mg/day on a 28-day cycle. Dose increments between cohorts will not exceed 100% of the dose in previous cohort. Patients in Part B will be treated with a schedule of 4d on/24d off (Q4W) at the Maximum tolerated dose (MTD) established from Part A.
  Interventions: Drug: CC-95775

INTERVENTIONS:
Drug: CC-95775 — CC-95775

SUMMARY:
CC-95775-ST-001 is an open-label, Phase 1B, dose escalation and expansion study of CC-95775 in subjects with advanced or unresectable solid tumors, including laBCC, and relapsed/ refractory non-Hodgkin's lymphoma (NHL). The dose escalation part (Part A) of the study will explore escalating oral doses of CC-95775 administered on a 4d on/24d off schedule to estimate the MTD of CC-95775. A mTPI-2 will help guide CC-95775 dose escalation decisions with the final decisions made by an SRC. Approximately 20 subjects will be enrolled.

The expansion cohort (Part B) will evaluate the safety, PK, PD safety and preliminary activity of CC-95775 in advanced solid tumors, including laBCC. Approximately 20 subjects will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the criteria below to be enrolled in dose escalation (Part A) and in dose expansion (Part B) of this study.

1. Men and women ≥ 18 years of age, at the time of signing the ICF.
2. Subject must understand and voluntarily sign an ICF prior to any study-specific assessments/procedures being conducted.
3. Subject is willing and able to adhere to the study visit schedule and other protocol requirements.
4. Subjects with histological or cytological confirmation of either:

   Advanced or unresectable ST, laBCC or R/R NHL.
   * Subjects with solid tumors including those who have progressed on (or not been able to tolerate due to medical comorbidities or unacceptable toxicity) standard anticancer therapy or for whom no other approved conventional therapy exists.
   * Subjects with laBCC must have unresectable disease which must have progressed after treatment with a smoothened inhibitor (SMOi) or who are intolerant of SMOi on (or not been able to tolerate due to medical comorbidities or unacceptable toxicity).
   * For relapsed/ refractory NHL following at least 2 prior lines of therapy (e.g. subjects have failed at least one line of standard therapy and have received at least one prior line of salvage therapy) OR have failed at least one prior line of standard therapy and are not eligible for autologous stem cell transplant (ASCT) OR have declined ASCT; transformed lymphoma following chemotherapy for lower grade lymphoma and at least one standard treatment regimen for DLBCL.

     * Subjects with two or more lines of systemic therapy who have been treated with and have lack of response or have responded and relapsed after chimeric antigen receptor T-cell (CAR-T) therapy, if such therapy is available, OR are ineligible for CAR-T therapy at the time of enrollment, OR declined CAR-T therapy.

   Subjects must have at least one site of measurable disease according to RECIST 1.1 Previously irradiated lesions are not considered evaluable; for subjects with R/R NHL, bi-dimensionally measurable disease on cross sectional imaging by CT or MRI, with at least one lesion >1.5 cm in its greatest transverse diameter, as defined by the IWG criteria. For subjects with rare malignancies, not falling into the above categories and who might benefit from a treatment with BET inhibitor, evaluable disease can be considered.
5. Subjects consent to tumor archive material analysis. Tumor biopsies to be collected whenever safe and feasible will be collected in Part A. Subjects consents to mandatory tumor biopsies (Screening and on treatment) in Part B.
6. ECOG PS of 0 to 1.
7. Subjects must have the following laboratory values at Screening:

   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L without growth factor support for 7 days (14 days if subject received peg-filgrastim).
   * Hemoglobin (HGB ≥10 g/dL (≥ 8g/dL for DLBCL subjects).
   * Platelet count (PLT) ≥150 x 109/L (≥100 x 109/L without transfusion for 7 days for DLBCL subjects).
   * Serum potassium concentration within normal range, or correctable with supplements
   * Serum glutamic oxaloacetic transaminase (SGOT)/aspartate aminotransferase (AST) and serum glutamate pyruvic transaminase (SGPT)/alanine aminotransferase (ALT) ≤ 3.0 x Upper Limit of Normal (ULN).
   * Serum total bilirubin ≤ 1.5 x ULN.
   * Serum creatinine ≤ 1.5 x ULN or measured glomerular filtration rate (GFR) ≥ 50 mL/min/1.73 m2 using an exogenous filtration marker such as iohexol, inulin, 51Cr EDTA or 1125 iothalamate, or creatinine clearance of ≥ 50 mL/min using Cockroft-Gault equation.
   * Subjects must have serum albumin > 3.5 g/dL.
   * PT (or INR) and APTT within normal range.
8. Subjects must agree not to share study drugs with another person
9. Females of childbearing potential

   * A female of childbearing potential (FCBP) is a female who: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy, or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy or other medical condition does not rule out childbearing potential) for at least 12 consecutive months and verified by an FSH blood test at screening.
   * FCBP must either commit to true abstinence from heterosexual intercourse (which must be reviewed monthly and source documented) or to use one highly effective contraceptive method plus one barrier method. True abstinence is acceptable when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception). Highly effective contraceptive methods are combined (containing estrogen and progestogen) or progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, intravaginal, patch, or implantable); bilateral tubal ligation; intrauterine device; intrauterine hormone-releasing system; or vasectomized partner sterilization (note that vasectomized partner is a highly effective birth control method provided that partner is the sole sexual partner of the FCBP trial participant and that the vasectomized partner has received medical assessment of the surgical success). Barrier methods are male or female latex or synthetic condom, diaphragm, cervical cap or sponge with spermicide, barrier contraceptive with spermicide. These measures should be used from signing the ICF, throughout the study, and for up to 44 days following the last dose of CC-95775.
   * Have two negative pregnancy tests as verified by the investigator prior to starting CC-95775.
   * Pregnancy testing:
   * A negative serum pregnancy test (or β-subunit of human chorionic gonadotropin (β-hCG pregnancy test) at Screening verified by the Investigator.
   * A negative serum or urine pregnancy test (or β-subunit of human chorionic gonadotropin (β-hCG pregnancy test) on Day 1 of dosing verified by the Investigator prior to dosing.
   * Agree to ongoing pregnancy testing during the course of the study, and after the end of study treatment. This applies even if the subject practices true abstinence from heterosexual contact.
10. Male subjects must practice true abstinence (which must be reviewed on a monthly basis) or agree to use a condom (a latex or non-latex synthetic condom is required) during sexual contact with a pregnant female or a FCBP and will avoid conceiving from signing the ICF, while participating in the study, during dose interruptions, and for at least 104 days following CC-95775 discontinuation, even if he has undergone a successful vasectomy. True abstinence is acceptable when this is in line with the preferred and usual lifestyle of the subject [female partner's periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception].

    * Males must agree not to donate semen or sperm for at least 104 days following CC-95775 discontinuation.
    * Other than the subject, FCBP and males able to father a child should not handle the study drugs or touch the capsules, unless gloves are worn.

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment (in Part A and Part B):

1. Subject has received anti-cancer therapy (either approved or investigational) within ≤ 4 weeks or 5 half-lives, whichever is shorter, prior to starting CC-95775.

   • < 42 days for prior nitrosureas or mitomycin C
2. Toxicities resulting from prior systemic cancer therapies must have resolved to ≤ NCI CTCAE Grade 1 prior to starting CC-95775 treatment (with exception of Grade 2 peripheral neuropathy and alopecia).
3. Subject has received autologous hematologic stem cell transplant (HSCT) ≤ 3 months prior to starting CC-95775 treatment. Subjects with allogeneic HSCT will not be allowed on this protocol.
4. Subject has undergone major surgery ≤ 4 weeks or minor surgery ≤ 2 weeks prior to starting CC-95775 or who have not recovered from surgery.
5. Subject has completed any radiation treatment < 4 weeks prior to starting CC-95775 (with exception of palliative bone radiotherapy for which 2-week period is required).
6. Subject has persistent diarrhea due to a malabsorptive syndrome (such as celiac sprue or inflammatory bowel disease) ≥ NCI CTCAE Grade 2, despite medical management, or any other significant GI disorder that could affect the absorption of CC-95775.
7. Subjects with symptomatic or uncontrolled ulcers (gastric or duodenal), particularly those with a history of and/or risk of perforation and GI tract hemorrhages.
8. Subjects with symptomatic or uncontrolled diabetes mellitus.
9. Symptomatic, untreated, or unstable central nervous system (CNS) metastases, (except in case of CNS primary tumors).

   * Subjects recently treated with whole brain radiation or stereotactic radiosurgery for CNS metastases must have completed therapy at least 4 weeks prior to starting CC-95775 and have a follow-up brain CT or MRI demonstrating either stable or improving metastases 4 or more weeks after completion of radiotherapy (the latter to be obtained as part of the Screening Assessments.
   * Subjects must be asymptomatic and off steroids or on stable dose of steroids for at least 4 weeks (<4 mg/day dexamethasone or equivalent) or on tapering dose of steroids.
10. Known symptomatic acute or chronic pancreatitis.
11. Impaired cardiac function or clinically significant cardiac diseases, including any of the following:

    * LVEF < 45% as determined by multiple gated acquisition scan (MUGA) or echocardiogram (ECHO).
    * Complete left bundle branch or bifascicular block.
    * Congenital long QT syndrome.
    * Persistent or clinically meaningful ventricular arrhythmias or atrial fibrillation.
    * QTcF ≥ 480 msec on Screening ECG (mean of triplicate recordings).
    * Unstable angina or myocardial infarction ≤ 6 months prior to starting CC-95770.
    * Other clinically significant heart disease such as congestive heart failure requiring treatment or uncontrolled hypertension (blood pressure ≥ 160/95 mm Hg).
12. Pregnant or nursing females.
13. Known HIV infection
14. Known chronic active hepatitis B or C virus (HBV, HCV) infection.

    * Subjects who are seropositive due to HBV vaccination are eligible.
    * Subjects who have no active viral infection and are under adequate prophylactics against HBV re-activation are eligible.
    * Subjects with HCC are exempt from the above criteria.
15. Ongoing treatment with chronic, therapeutic dosing of anti-coagulants (e.g., warfarin, low molecular weight heparin, Factor Xa inhibitors, thrombin antagonists). Low dose, low molecular weight heparin for catheter maintenance is allowed.
16. History of concurrent second cancers requiring active, ongoing systemic treatment.
17. Subjects with a history of clinically significant cognitive disorder(s) or active cognitive disorder(s).
18. Evidence of history of bleeding diathesis. Any hemorrhage/bleeding event > CTCAE Grade 2 or hemoptysis > 1 teaspoon within 4 weeks prior to the first dose
19. Subject has any significant medical condition (e.g., active or uncontrolled infection or renal disease), laboratory abnormality, or psychiatric illness that would prevent the subject from participating (or compromise compliance) in the study or would place the subject at unacceptable risk if he/she were to participate in the study.
20. Subject has any condition that confounds the ability to interpret data from the study.
21. Subjects with poor bone marrow reserve as assessed by the Investigator such as in the following conditions:

    * Having received extensive bone radiotherapy
    * Having experienced several episodes of bone marrow aplasia in previous treatments
    * Confirmed histological bone marrow cancer infiltration (with exemption of NHL)
    * Requiring regular hematopoietic support (blood transfusion, erythropoietin, G-CSF)
22. Subjects with severely compromised pulmonary function and/or requiring chronic oxygen administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-10-24 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2021-10-25 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | C1 Up to approximately 28 days
  is defined as any toxicities occurring within the DLT assessment unless the event can clearly be determined to be unrelated to CC-95775.
Maximum Tolerated Dose (MTD) | Part A of the study- estimated 12 months
  dose level that could be given such that the estimated DLT probability is closest to 25%.
Non-tolerated Dose (NTD) | Part A of the study-estimated 12 months
  The dose that is higher than MTD
Adverse Events (AEs) | From signature of the informed consent until at least 28 days after the last dose of study treatment
  Number of participants with adverse event. An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a subject during the course of a study

SECONDARY OUTCOMES:
Pharmacokinetics - Cmax of CC-95775 | Part A and part B of the study, estimated 24 months total
  Maximum plasma concentration of drug
Pharmacokinetics - AUC of CC-95775 | Part A and part B of the study, estimated 24 months total
  Area under the curve
Pharmacokinetics - Tmax of CC-95775 | Part A and part B of the study, estimated 24 months total
  Time to peak plasma concentration
Pharmacokinetics - t1/2 of CC-95775 | Part A and part B of the study, estimated 24 months total
  Half-life the time it takes for the concentration of the drug in the plasma to be reduced by 50%
Pharmacokinetics - CL/F of CC-95775 | Part A and part B of the study, estimated 24 months
  Measurement of the volume of plasma from which a substance is completely removed per unit time
Pharmacokinetics - Vz/F of CC-95775 | Part A and part B of the study, estimated 24 months
  Apparent volume of distribution. It is the volume needed to account for the total amount of drug in the body if the drug was evenly distributed throughout the body and in the same concentration as the site of sample collection such as peripheral venous plasma
Evaluate the pharmacodynamic (PD) effects of CC-95775 on gene expression in peripheral blood and in tumor tissue. | Part B of the study, estimated 12 months
  Changes in the expression of genes associated to BET inhibitors in PBMCs and/or other genes, such as GLI1, MYC, in tumor biopsy may provide confirmation that a dose is pharmacologically active and enable identification of dose, which results in optimal target engagement

CONTACTS AND LOCATIONS:
Overall Officials: Pilar Lardelli, MD PhD, Study Director — Celgene
Locations (5):
- France (3):
  - Institut Curie, Paris
  - Hopital Saint Louis, Paris
  - Centre Eugene Marquis, Rennes
- Spain (2):
  - Hospital de Madrid Norte- Sanchinarro, Madrid
  - Clinica Universidad de Navarra, Pamplona

IPD SHARING:
Plan to Share IPD: Yes
https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/